CLINICAL TRIAL: NCT01636076
Title: A Randomized, Double-blind, 12-week Treatment, Parallel-group Study to Evaluate the Efficacy and Safety of QMF149 (150 µg/160 µg o.d.) Compared With Salmeterol Xinafoate/Fluticasone Propionate (50 µg/500 µg b.i.d.) in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy and Safety of QMF149 vs. Salmeterol Xinafoate/Fluticasone Propionate in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQMF149F2202; 2012-001172-12 (EudraCT Number)
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: COPD
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — QMF149; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- QMF149 (Experimental): QMF149 (Indacaterol acetate/Mometasone furoate) 150/160 µg o.d. delivered via Concept1 device
  Interventions: Drug: QMF149
- Salmeterol xinafoate/fluticasone propionate (Active Comparator): Salmeterol xinafoate/fluticasone propionate 50/500 µg b.i.d, delivered via Accuhaler®
  Interventions: Drug: Salmeterol

INTERVENTIONS:
Drug: QMF149 — delivered via Concept1 device
  Arms: QMF149
Drug: Salmeterol — delivered via Accuhaler®
  Arms: Salmeterol xinafoate/fluticasone propionate

SUMMARY:
To compare the efficacy, safety and pharmacokinetics of QMF149 delivered via Concept1 to salmeterol xinafoate/fluticasone propionate delivered via Accuhaler in adult patients with COPD

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to very severe COPD (GOLD 2 to GOLD 4) according to the 2011 Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines
* Patients with a post-bronchodilator FEV1 < 70% of the predicted normal, and a post-bronchodilator FEV1/FVC < 0.70 at run-in (Visit 101).
* Current or ex-smokers who have a smoking history of at least 10 pack years (defined as the number of packs of 20 cigarettes smoked per day multiplied by number of years the patient smoked. e.g.10 pack years = 1 pack /day x 10 yrs, or ½ pack/day x 20 yrs). An ex-smoker may be defined as a subject who has not smoked for ≥ 6 months at screening.

Exclusion Criteria:

* Patients who have had a COPD exacerbation that required treatment with antibiotics and/or oral corticosteroids and/or hospitalization in the 6 weeks prior to screening (Visit 1).
* Patients who develop a COPD exacerbation between screening (Visit 1) and treatment (Visit 201) will not be eligible but will be permitted to be re-screened after a minimum of 6 weeks after the resolution of the COPD exacerbation.
* Patients who have had a respiratory tract infection within 4 weeks prior to screening Visit 1.
* Patients who develop a respiratory tract infection between screening (Visit 1) and treatment (Visit 201) will not be eligible, but will be permitted to be re-screened 4 weeks after the resolution of the respiratory tract infection.
* Patients requiring long term oxygen therapy prescribed for >12 hours per day.
* Patients with, a) any history of asthma or, b) onset of respiratory symptoms prior to age 40 years.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 629 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (98):
- Australia (11):
  - Novartis Investigative Site, Concord, New South Wales
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, New Lambton Heights, New South Wales
  - Novartis Investigative Site, Redcliffe, Queensland
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Daw Park, South Australia
  - Novartis Investigative Site, Woodville South, South Australia
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, Fitzroy, Victoria
  - Novartis Investigative Site, Franston, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Halen
  - Novartis Investigative Site, Liège
- Bulgaria (6):
  - Novartis Investigative Site, Rousse, Bulgaria
  - Novartis Investigative Site, Varna, Bulgaria
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Stara Zagora
  - Novartis Investigative Site, Veliko Tarnovo
- Denmark (4):
  - Novartis Investigative Site, Hellerup, Denmark
  - Novartis Investigative Site, Hvidovre, Denmark
  - Novartis Investigative Site, Copenhagen NV
  - Novartis Investigative Site, Odense C
- Finland (3):
  - Novartis Investigative Site, Turku, Finland
  - Novartis Investigative Site, Pori
  - Novartis Investigative Site, Tampere
- Germany (10):
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Wiesbaden, Germany
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Donaustauf
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Witten
- Greece (6):
  - Novartis Investigative Site, Heraklion Crete, Crete
  - Novartis Investigative Site, Athens, Greece
  - Novartis Investigative Site, Larissa, Greece
  - Novartis Investigative Site, Thessaloniki, Greece
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Athens - GR
- Hong Kong (2):
  - Novartis Investigative Site, Hong Kong, Hong Kong
  - Novartis Investigative Site, New Territories, Hong Kong
- Hungary (10):
  - Novartis Investigative Site, Budapest, Hungary
  - Novartis Investigative Site, Nyíregyháza, Hungary
  - Novartis Investigative Site, Szarvas, Hungary
  - Novartis Investigative Site, Balasagyarmat
  - Novartis Investigative Site, Farkasgyepű
  - Novartis Investigative Site, Kapuvár
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Siófok
  - Novartis Investigative Site, Sopron
  - Novartis Investigative Site, Veszprém
- Israel (7):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv
- Malaysia (3):
  - Novartis Investigative Site, Batu Caves
  - Novartis Investigative Site, Kuala Lumpur
  - Novartis Investigative Site, Taiping
- Poland (11):
  - Novartis Investigative Site, Gdansk, Poland
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Iława
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Ostrów Wielkopolski
  - Novartis Investigative Site, Piła
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Szczecin
  - Novartis Investigative Site, Tarnów
  - Novartis Investigative Site, Wroclaw
- Romania (4):
  - Novartis Investigative Site, Constanța, Jud. Constanta
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Târgu Mureş
- Novartis Investigative Site, Singapore, Singapore, Singapore
- South Africa (5):
  - Novartis Investigative Site, Johannesburg, Gauteng
  - Novartis Investigative Site, Durban, South Africa
  - Novartis Investigative Site, Bloemfontein
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, eMkhomazi
- Spain (3):
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
- Sweden (4):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Vällingby
- Thailand (5):
  - Novartis Investigative Site, Taladkwan, Changwat Nonthaburi
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Muang
  - Novartis Investigative Site, Nakhon Naiyok
  - Novartis Investigative Site, Songkhla

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Started | 316 | 313
Completed | 299 | 288
Not Completed | 17 | 25
Not completed — Terminated by sponsor | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Non-compliance with study treatment | 1 | 1
Not completed — Adverse Event | 6 | 11
Not completed — Withdrawal by Subject | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate | Total
Number analyzed (Participants) | 316 | 313 | 629
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (7.74) | 64.1 (7.89) | 64.5 (7.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 86 | 169
  Male | 233 | 227 | 460
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 32 | 30 | 62
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 273 | 276 | 549
  Other | 9 | 6 | 15
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mixed Model for Repeated Measures (MMRM): Between-treatment Comparisons for Trough FEV1 (L) on Day 85
Description: Spirometry is conducted according to the global standard. Trough FEV1 is defined as the average of the 23 hour 10 minute and 23 hour 45 minute post dose FEV1 readings.
Time Frame: 12 weeks
Population: All randomized patients were included in the Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 316 | 313
Liters
  Full analysis set (n=291,282) | 1.270 (0.0124) | 1.215 (0.0124)
  Per protocol set (n=259,251) | 1.277 (0.0136) | 1.228 (0.0137)

2. Secondary Outcome: Trough FEV1 After First Dose and After 4 Weeks of Treatment
Description: Spirometry is conducted according to the global standard. FEV1 is measured at pre-dose and post dose up to 1 hours on Day 1 and Day 28; 24 hours post-dose on Day 29 and 85. In a subset of approximately 60 patients, FEV1 is measured up to 20 hours postdose on Day 28 and Day 84.
Time Frame: Day 1 and Day 85
Population: All randomized patients were included in the Safety analysis set (SAF) and Full analysis set (FAS).
Measure: Mean (Standard Error); unit: Liters
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 316 | 313
Liters
  Baseline Day 2 (n=286, 302) | 1.147 (0.0237) | 1.167 (0.0264)
  Day 2 (n=286, 302) | 1.216 (0.0106) | 1.243 (0.0104)
  Baseline Day 29 (n=293, 296) | 1.148 (0.0236) | 1.178 (0.0266)
  Day 29 (n=293,296) | 1.277 (0.0119) | 1.247 (0.0119)
  Day 84 baseline (n=289,287) | 1.144 (0.0240) | 1.187 (0.0267)
  Day 84 (n=289,287) | 1.269 (0.0139) | 1.208 (0.0139)

3. Secondary Outcome: Mixed Model for Repeated Measures (MMRM): Between-treatment Comparisons for FEV1 (L), by Visit and Timepoint
Time Frame: Day 1 through day 85
Population: Full analysis set consisting of all randomized patients
Measure: Least Squares Mean (Standard Error); unit: liter
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 316 | 313
liter
  Absolute Value Day 1/5min (n=290,298) | 1.254 (0.0069) | 1.198 (0.0068)
  Absolute Value Day 1/30 min (n=294,306) | 1.281 (0.0079) | 1.250 (0.0087)
  Absolute Value Day 1/60min (n=300,303) | 1.281 (0.0087) | 1.256 (0.0087)
  Absolute Value Day 2/ 23 hr 10 min (n=288,295) | 1.213 (0.0108) | 1.239 (0.0107)
  Absolute Value Day 2/ 23 hr 45 min (n=297,305) | 1.215 (0.0106) | 1.244 (0.0105)
  Absolute Value Day 28/ -50min (n=288,295) | 1.265 (0.0132) | 1.287 (0.0139)
  Absolute Value Day 28/ -15min (n=292,290) | 1.287 (0.0132) | 1.235 (0.0140)
  Absolute Value Day 28/ 5min (n=290,289) | 1.329 (0.0113) | 1.268 (0.0113)
  Absolute Value Day 28/ 30min (n=293,290) | 1.352 (0.0118) | 1.298 (0.0118)
  Absolute Value Day 28/ 60min (n=292,290) | 1.353 (0.0123) | 1.298 (0.0122)
  Absolute Value Day 29/ 23 hr 10 min (n=285,292) | 1.269 (0.0118) | 1.242 (0.0117)
  Absolute Value Day 29/ 23 hr 45 min (n=290,295) | 1.281 (0.0123) | 1.254 (0.0122)
  Absolute Value Day 84/ -50 min (n=286,278) | 1.259 (0.0140) | 1.195 (0.0141)
  Absolute Value Day 84/ -15 min (n=282,285) | 1.282 (0.0146) | 1.222 (0.0147)
  Absolute Value Day 84/ 5 min (n=280,279) | 1.336 (0.0128) | 1.243 (0.0128)
  Absolute Value Day 84/ 30 min (n=286,280) | 1.352 (0.0124) | 1.277 (0.0124)
  Absolute Value Day 84/ 60 min (n=287,281) | 1.351 (0.0128) | 1.283 (0.0128)
  Absolute Value Day 84/ 23 hr 10 min (n=292,291) | 1.264 (0.0125) | 1.212 (0.0125)
  Absolute Value Day 84/ 23 hr 45 min (n=291,285) | 1.273 (0.0125) | 1.221 (0.0126)

4. Secondary Outcome: Forced Vital Capacity (FVC) at Each Timepoint
Description: Spirometry is conducted according to the global standard. FVC is measured at pre-dose and post dose up to 4 hour on Day 1, Day 28, and Day 84, at post dose 12 hour, 23 hour 10 minute and 23 hour 45 minutes on Day 2 and Day 29, and at pre-dose 50 min and 15 min on Day 2, Day 28, and Day 84.
Time Frame: Day 1, Day 2, Day 28, Day , Day 29, Day 84, Day 85
Population: Full analysis set consisting of all randomized patients
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 316 | 313
liters
  Baseline (n=316,313) | 2.460 (0.6969) | 2.481 (0.7209)
  Day 1/ 5 min (n=299,298) Change | 0.179 (0.2165) | 0.060 (0.1404)
  Day 1/ 30 min (n=302,306) Change | 0.207 (0.2279) | 0.129 (0.1953)
  Day 1/ 60 min (n=308,303) Change | 0.222 (0.2472) | 0.152 (0.2287)
  Day 1/ 4 hr (n=302,297) Change | 0.217 (0.2847) | 0.183 (0.2611)
  Day 2/ 23hr 10 min (n=297,296) Change | 0.089 (0.2518) | 0.092 (0.2896)
  Day 2/ 23hr 45 min (n=307,306) Change | 0.083 (0.2583) | 0.092 (0.2815)
  Day 28 / -50 min (n=295,296) Change | 0.132 (0.2806) | 0.068 (0.2814)
  Day 28 / -15 min (n=300,291) Change | 0.161 (0.3090) | 0.072 (0.2892)
  Day 28 / 5 min (n=297,290) Change | 0.238 (0.3163) | 0.122 (0.3068)
  Day 28 / 30 min (n=301,291) Change | 0.263 (0.3169) | 0.168 (0.3166)
  Day 28 / 60 min (n=299,292) Change | 0.279 (0.3261) | 0.189 (0.3350)
  Day 29 / 23hr 10 min (n=293,293) Change | 0.121 (0.2955) | 0.084 (0.2817)
  Day 29 /23hr 45 min (n=299,296) Change | 0.133 (0.3132) | 0.097 (0.2965)
  Day 84 / -50min (n=295,279) Change | 0.125 (0.2979) | 0.144 (0.3570)
  Day 84 /-15 min (n=291,286) Change | 0.144 (0.3234) | 0.049 (0.3519)
  Day 84 / 5 min (n=288,290) Change | 0.229 (0.3370) | 0.076 (0.3729)
  Day 84 /30 min (n=295,281) Change | 0.255 (0.3344) | 0.120 (0.3537)
  Day 84 / 60 min (n=296,282) Change | 0.272 (0.3295) | 0.159 (0.3648)
  Day 85 / 23 hr 10 min (n=302,292) Change | 0.113 (0.3132) | 0.022 (0.3482)
  Day 85 / 23 hr 45 min (n=301,286) Change | 0.126 (0.3206) | 0.035 (0.3620)

5. Secondary Outcome: FEV1/FVC at Each Timepoint
Description: Spirometry is conducted according to the global standard. FEV1/FVC is measured at pre-dose and post dose up to 4 hour on Day 1, Day 28, and Day 84, at post dose 12 hour, 23 hour 10 minute and 23 hour 45 minutes on Day 2 and Day 29, and at pre-dose 50 min and 15 min on Day 2, Day 28, and Day 84.
Time Frame: Day 1, Day 2, Day 28, Day , Day 29, Day 84, Day 85
Population: Full analysis set consisting of all randomized patients
Measure: Mean (Standard Deviation); unit: FEV1/ FVC (%)
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 316 | 313
FEV1/ FVC (%)
  Baseline (n=316, 313) | 46.786 (10.0306) | 46.859 (10.0392)
  Day 1 / 5 min (n=299, 298) change | 0.488 (2.9633) | 0.047 (2.1366)
  Day 1 / 30 min (n=302,306) change | 0.955 (3.0166) | 0.879 (2.7281)
  Day 1 / 60 min (n=308,303) change | 1.112 (3.1413) | 1.182 (3.0612)
  Day 1 / 4 hr (n=302, 297) change | 1.045 (3.3917) | 1.397 (3.2407)
  Day 2 / 23 Hr 10 min (n=297,296) change | 0.503 (3.3450) | 1.042 (3.2074)
  Day 2 / 23 Hr 45 min (n=307,306) change | 0.583 (3.4552) | 1.319 (3.1977)
  Day 28 / -50 min (n=295,296) change | 1.463 (3.7864) | 1.140 (3.8900)
  Day 28 / -15 min (n=300,291) change | 1.837 (3.9769) | 1.495 (3.7597)
  Day 28 / 5 min (n=297,290) change | 1.951 (4.0512) | 1.581 (4.006)
  Day 28 / 30 min (n=301,291) change | 2.296 (4.4904) | 1.873 (4.2723)
  Day 28 / 60 min (n=299,292) change | 2.525 (4.3228) | 2.060 (4.4398)
  Day 28 / 4 hr (n=44,45) change | 4.034 (5.2622) | 2.322 (4.0257)
  Day 28 / 11hr 10 min (n=47,44) change | 2.553 (4.0260) | 1.909 (3.9389)
  Day 28 / 11hr 45 min (n=43,42) change | 2.791 (4.1708) | 2.476 (4.3978)
  Day 28 / 16 hr (n=40,41) change | 2.250 (3.4006) | 2.305 (4.3111)
  Day 28 / 20 hr (n=43,44) change | 2.535 (3.5379) | 2.250 (3.9935)
  Day 29 / 23 hr 10 min (n=293,293) change | 1.771 (4.0730) | 1.319 (3.8200)
  Day 29 / 23 hr 45 min (n=299,296) change | 2.000 (4.0562) | 1.566 (3.9704)
  Day 84 / -50 min (n=295,279) change | 1.449 (4.1145) | 1.068 (4.1776)
  Day 84 / -15 min (n=291,286) change | 2.155 (4.0673) | 1.584 (4.3278)
  Day 84 / 5 min (n=288,280) change | 2.332 (4.1032) | 1.796 (4.2310)
  Day 84 / 30 min (n=295,281) change | 2.420 (4.3561) | 2.062 (4.3941)
  Day 84 / 60 min (n=296,282) change | 2.571 (4.4128) | 2.067 (4.3512)
  Day 84 / 4 hr (n=45,44) change | 2.389 (3.7079) | 2.682 (4.3269)
  Day 84 / 11hr 10 min (n=45,43) change | 1.944 (4.0833) | 2.105 (3.8754)
  Day 84 / 11 hr 45 min (n=39,39) change | 2.538 (3.7895) | 2.295 (4.1147)
  Day 84 / 16 hr (n=41,39) change | 1.415 (4.0588) | 1.962 (3.6981)
  Day 84 / 20 hr (n=44,43) change | 2.364 (4.4315) | 1.837 (3.7713)
  Day 84 / 23 hr 10 min (n=302,292) change | 1.856 (4.4315) | 1.414 (4.0356)
  Day 84 / 23 hr 45 min (n=301,286) change | 2.098 (4.3676) | 1.593 (4.2110)

6. Secondary Outcome: FEV1 (L) on Day 1 Between-treatment Comparisons of AUC (5min - 4h)
Description: Spirometry is conducted according to the global standard. FEV1 AUC (5 min-4 h), Scheduled (not actual) time points are to be used. The standardized AUC(5 min - 4 h) for FEV1 will be summarized by treatment.
Time Frame: Day 1
Population: Full analysis set consisting of all randomized patients
Measure: Least Squares Mean (Standard Error); unit: Liters * hours
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 316 | 313
Liters * hours
  Day 1 baseline (n=303,311) | 1.142 (0.0233) | 1.169 (0.0259)
  Day 1 post (n=303,311) | 1.277 (0.0086) | 1.260 (0.0085)

7. Secondary Outcome: FEV1 AUC (5 Min-4 h),
Description: Spirometry is conducted according to the global standard. FEV1 AUC (5 min-4 h), (5 min-24 h) is measured after the first dose on Day 1 and on Day 28 and Day 84 in a subset of approximately 60 patients. Scheduled (not actual) time points are to be used. The interpretation of FEV1 at time 0 is the baseline value at the randomization visit and the latest pre-dose value (-50 min or -15 min) at subsequent visits. The standardized AUC(5 min - 4 h) for FEV1 will be summarized by treatment. The same will be repeated for standardized AUC for FEV1 between 5 min and 24 hours post morning dose.
Time Frame: Day 1(Baseline), Day 28, Day 84
Population: 24 hr profiling subgroup
Measure: Least Squares Mean (Standard Error); unit: Liters*hours
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 50 | 50
Liters*hours
  Day 1 baseline (n=46,47) | 1.302 (0.0278) | 1.331 (0.0282)
  Day 28 (n=45,46) | 1.410 (0.0353) | 1.355 (0.0355)
  Day 84 (n=44,46) | 1.387 (0.0401) | 1.372 (0.0401)

8. Secondary Outcome: Mixed Model for Repeated Measures (MMRM): Between-treatment Comparisons for AUC (5 Min - 23 h 45 Min) for FEV1 (L) on Day 28 and Day 84 (Full Analysis Set, 24-h Profiling Subgroup)
Description: as for outcome 7
Time Frame: Day 28, Day 84
Population: Peak FEV1 was calculated for all subjects in the FAS at Day 1 (Visit 201) and was calculated for all subjects in the 24-h profiling subset of the FAS at Day 1 (Visit 201), Day 28 (Visit 203) and Day 84 (Visit 205).
Measure: Least Squares Mean (Standard Error); unit: Liters*hours
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 50 | 50
Liters*hours
  Day 28 (n=45,46) | 1.352 (0.0428) | 1.298 (0.0431)
  Day 85 (n=47,47) | 1.317 (0.0454) | 1.303 (0.0459)

9. Secondary Outcome: The Usage of Rescue Medication (Short Acting β2-agonist)
Description: Participants record the number of puffs of rescue medication taken in the previous 12 hours each morning and evening throughout the 12 week treatment period.
Time Frame: 12 weeks
Population: Full analysis set consisting of all randomized patients
Measure: Least Squares Mean (Standard Error); unit: Number of puffs
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 316 | 313
Number of puffs
  Daily Change Weeks 1-12 (n-281,274) | -1.064 (0.1615) | -0.593 (0.1621)
  Daytime Change Weeks 1-12 (n=276-272) | -0.625 (0.1021) | -0.300 (0.1026)
  Nighttime Change Weeks 1-12 (n=281,271) | -0.452 (0.0748) | -0.308 (0.0751)

10. Secondary Outcome: The Overall Change in Usage of Rescue Medication (Short Acting β2-agonist) .
Description: This value represents the percent of days in the study where no rescue medication was needed.
Time Frame: Baseline to 12 weeks
Population: Full analysis set consisting of all randomized patients
Measure: Least Squares Mean (Standard Error); unit: % of days
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 316 | 313
% of days | 8.796 (2.3845) | 2.538 (2.3980)

11. Secondary Outcome: Patient Reported Outcome Measures: SGRQ (St. George's Respiratory Questionnaire)
Description: A Total and three component scores are calculated: Symptoms; Activity; Impacts. Each component of the questionnaire is scored separately:The score for each component is calculated separately by dividing the summed weights by the maximum possible weight for that component and expressing the result as a percentage: Score = 100 x Summed weights from all positive items in that component divided by Sum of weights for all items in that component The Total score is calculated in similar way: Score = 100 x Summed weights from all positive items in the questionnaire divided by Sum of weights for all items in the questionnaire Sum of maximum possible weights for each component and Total: Symptoms 566.2 Activity 982.9 Impacts 1652.8 Total (sum of maximum for all three components) 3201.9 The proportion of patients who achieve a clinically important improvement of at least 4 units in the total SGRQ will be analyzed. The higher the score the more symptoms of disease are present.
Time Frame: 4 and 12 weeks
Population: Full analysis set : At baseline all subjects with a baseline value are included. At each post-baseline day, only subjects with a value at both baseline and the respective day are included. Baseline SGRQ was completed on Day 1 prior to first dose.
Measure: Mean (Standard Deviation); unit: Total Score
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 316 | 313
Total Score
  Baseline (n=314, 308) | 43.05 (18.515) | 42.28 (17.941)
  Day 28 Baseline (n=304,295) | 42.87 (18.392) | 42.47 (18.051)
  Day 28 Post (n=304,295) | 40.95 (18.527) | 42.18 (18.101)
  Day 28 Change (n=304,295) | -1.92 (11.383) | -0.29 (12.145)
  Day 84 Baseline (n=297,284) | 42.57 (18.322) | 42.03 (18.099)
  Day 84 Post (n=297,284) | 39.81 (19.057) | 41.01 (18.553)
  Day 84 Change (n=297,284) | -2.76 (13.062) | -1.02 (12.178)

12. Secondary Outcome: Analysis of the Proportion of Subjects With a Clinically Important Improvement of >=1 Point in the TDI (Transitional Dyspnoea Index)Focal Score by Visit
Description: A TDI focal score of ≥1 is considered to be a clinically important improvement from baseline. Analysis of the proportion of subjects with a clinically important improvement of >=1 point in the TDI focal score, by visit
Time Frame: 4 and 12 weeks
Population: Full analysis set, All randomized patients. When data were missing or insufficient for any one of the domains a focal score could not be calculated.
Measure: Number; unit: (%) showing clinical improvement
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 316 | 313
(%) showing clinical improvement
  Day 28 Change from baseline (n=291,294) | 43.3 (0.1314) [0.79 to 1.68] | 40.5 (0.1331)
  Day 84 Change from baseline (n=287,283) | 52.6 (0.1330) [0.99 to 2.05] | 45.9 (0.1390)

13. Secondary Outcome: Patient Reported Outcome Measures: COPD Assessment Test
Description: It consists of eight items, each presented as a semantic 6-point differential scale, providing a total score out of 40. A higher score indicates a worse health status. Scores of 0 - 10, 11 - 20, 21 - 30 and 31 - 40 represent a mild, moderate, severe or very severe clinical impact of COPD upon the patient.
Time Frame: Baseline, 4 and 12 weeks
Population: Full analysis set consisting of all randomized patients
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 316 | 313
Units on a scale
  Baseline (n= 311,308) | 16.3 (7.60) | 16.2 (7.48)
  Day 28 baseline (n=303,298) | 16.2 (7.58) | 16.2 (7.48)
  Day 28 Post (n=303,298) | 15.8 (7.63) | 16.8 (7.75)
  Day 28 Change (n=303,298) | -0.4 (5.56) | 0.6 (4.94)
  Day 84 Baseline (n=295,285) | 15.9 (7.54) | 16.1 (8.38)
  Day 84 Post (n=295,285) | 15.5 (7.56) | 16.3 (8.38)
  Day 84 change (n=295,285) | -0.4 (5.77) | 0.2 (5.84)

14. Secondary Outcome: Patient Reported Outcome Measures: Medical Outcome Study (MOS) Sleep Scale: Without Quantity Subscale
Description: Scoring the MOS Sleep Survey is a two-step process:• All items are scored so that a high score reflects more of the attribute implied by the scale name. Each item is converted to a 0 to 100 possible range so that the lowest and highest possible scores are set at 0 and 100, respectively. In this format, scores represent the achieved percentage of the total possible score. For example, a score of 50 represents 50% of the highest possible score.
  • Second, items within each scale are averaged together to create the 7 scale scores. Scales with at least one item answered can be used to generate a scale score. Items that are left blank (missing data) are not taken into account when calculating the scale scores. Scores represent the average for all items in the scale that the respondent answered. An additional measure is based on the average number of hours sleep each night during the past 4 weeks and are described in outcome measure 15.
Time Frame: Baseline, 4 and 12 weeks
Population: Full analysis set.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 302 | 296
Units on a scale
  Sleep disturbance Day 28 Baseline (n=290,285) | 49.6833 (8.57069) | 49.7616 (8.49307)
  Sleep disturbance Baseline (n=299,295) | 49.6423 (8.50059) | 49.9292 (8.51330)
  Sleep disturbance Day 28 post (n=290,285) | 50.9323 (8.92540) | 50.0858 (8.77110)
  Sleep disturbance Day 28 change (n=290,285) | 1.2490 (5.67591) | 0.3242 (6.63156)
  Sleep disturbance Day 84 Baseline (n=283,274) | 49.7622 (8.61100) | 49.6634 (8.41228)
  Sleep disturbance Day 84 Post (n=283,274) | 50.7508 (9.22016) | 50.2380 (9.07204)
  Sleep disturbance Day 84 Change (n=283,274) | 0.9887 (6.52972) | 0.5745 (6.45362)
  Sleep snoring Baseline (n=299,295) | 48.8815 (9.32313) | 49.8895 (9.18885)
  Sleep snoring Day 28 Baseline (n=290,285) | 48.8234 (9.40239) | 49.7733 (9.23030)
  Sleep snoring Day 28 Post (n=290,285) | 49.3476 (9.37744) | 49.5067 (9.39012)
  Sleep snoring Day 28 change(n=290,285) | 0.5241 (6.70023) | -0.2667 (7.06825)
  Sleep snoring Day 84 Baseline (n=283,274) | 48.8414 (9.29113) | 49.6385 (9.19681)
  Sleep snoring Day 84 post (n=283,274) | 49.4591 (9.29113) | 49.6108 (9.51632)
  Sleep snoring Day 84 change (n=283,274) | 0.6177 (7.42456) | -0.0277 (8.266668)
  Sleep shortness of breath Baseline (n=302,295) | 44.5221 (13.28329) | 45.4259 (11.51560)
  Sleep shortness of breath D 28 Bseline(n=293,285) | 44.6348 (13.15710) | 45.3292 (11.48556)
  Sleep shortness of breath D 28 post (n=293,285) | 45.8814 (11.85664) | 45.5774 (11.65379)
  Sleep shortness of breath D 28 change (n=293,285) | 1.2466 (12.21272) | 0.2481 (11.44262)
  Sleep shortness of breath D 84 Bseline (n=287,274) | 44.8645 (12.99605) | 45.3180 (11.37006)
  Sleep shortness of breath D 84 post (n=287,274) | 45.7676 (13.20151) | 45.7049 (11.84910)
  Sleep shortness of breath D 84 change (n=287,274) | 0.9031 (12.11351) | 0.3870 (10.97093)
  Sleep adequacy baseline (n=300,295) | 54.9999 (9.85865) | 54.9725 (9.41704)
  Sleep adequacy baseline D 28 (n=291,285) | 55.0531 (9.80609) | 55.0679 (9.30955)
  Sleep adequacy Post D 28 (n=291,285) | 55.2032 (10.04281) | 54.8296 (10.21011)
  Sleep adequacy Change D 28 (n=291,285) | 0.1501 (9.83920) | -0.2383 (9.21250)
  Sleep adequacy baseline D 84 (n=284,274) | 55.2125 (9.81055) | 55.1084 (9.20723)
  Sleep adequacy Post D 84 (n=284,274) | 55.2467 (10.00283) | 54.5424 (9.96705)
  Sleep adequacy change D 84 (n=284,274) | 0.0342 (8.81793) | -0.5659 (8.57800)
  Sleep somnolence baseline (n=302,296) | 47.6646 (9.56376) | 49.1709 (9.56807)
  Sleep somnolence baseline D28 (n=290,285) | 47.8711 (9.48940) | 49.1092 (9.58808)
  Sleep somnolence post D28 (n=290,285) | 48.4429 (9.93046) | 48.6761 (10.17850)
  Sleep somnolence change D28 (n=290,285) | 0.5718 (7.91162) | -0.4331 (8.67719)
  Sleep somnolence baseline D84 (n=284,274) | 47.7821 (9.53639) | 48.9335 (9.55603)
  Sleep somnolence post D84 (n=284,274) | 48.2568 (10.36223) | 49.0461 (9.54132)
  Sleep somnolence change D84 (n=284,274) | 0.4747 (8.11292) | 0.1126 (7.83662)
  Sleep Problems Index 1 Baseline (n=300,295) | 50.4795 (9.72203) | 50.8382 (9.16082)
  Sleep Problems Index 1 Baseline D28 (n=290,285) | 50.6034 (9.67464) | 50.7911 (9.13425)
  Sleep Problems Index 1 Post D28 (n=290,285) | 51.4799 (9.86137) | 50.7836 (10.02742)
  Sleep Problems Index 1 Change D28 (n=290,285) | 0.8764 (7.03960) | -0.0074 (7.73909)
  Sleep Problems Index 1 Baseline D84 (n=284,274) | 50.7327 (9.64776) | 50.6951 (9.09626)
  Sleep Problems Index 1 Post D84 (n=284,274) | 51.3590 (10.16584) | 50.9888 (9.54642)
  Sleep Problems Index 1 Change D84 (n=284,274) | 0.6263 (7.22742) | 0.2938 (7.08082)
  Sleep Problems Index 2 baseline (n=299,295) | 50.4610 (9.14154) | 51.0701 (8.62899)
  Sleep Problems Index 2 baseline D 28 (n=289,285) | 50.5720 (9.15508) | 50.9923 (8.60656)
  Sleep Problems Index 2 Post D 28 (n=289,285) | 51.5578 (9.43365) | 51.0116 (9.33837)
  Sleep Problems Index 2 Change D 28 (n=289,285) | 0.9858 (6.00711) | 0.0193 (6.99119)
  Sleep Problems Index 2 Baseline D 84 (n=283,274) | 50.6880 (9.16092) | 50.8848 (8.58893)
  Sleep Problems Index 2 Post D 84 (n=283,274) | 51.4615 (9.79518) | 51.1511 (9.09673)
  Sleep Problems Index 2 Change D 84 (n=283,274) | 0.7735 (6.66709) | 0.2663 (6.29393)

15. Secondary Outcome: Patient Reported Outcome Measures: Medical Outcome Study (MOS) Sleep Scale: Sleep Quantity Subscale
Description: The sleep quantity subscale,which refers to question 2 of the PRO: On average, how many hours did you sleep each night during the past 4 weeks. More hours of sleep indicate better outcome.
Time Frame: Baseline, 4 and 12 weeks
Population: Full analysis set.Higher scores show better outcomes.Excepting the sleep quantity subscale,scoring the MOS requires two steps:(a) assigning a point value to each response and (b) summing the point values for all the items in a given subscale or index. Each subscale and index score is then converted to a T score with a mean of 50 and an SD of 10.
Measure: Mean (Standard Deviation); unit: hours of sleep
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 302 | 296
hours of sleep
  Sleep quantity Baseline (n=301,295) | 6.5565 (1.44169) | 6.6203 (1.34895)
  Sleep quantity Baseline D28(n=292,285) | 6.5702 (1.44879) | 6.6351 (1.35775)
  Sleep quantity Post D28(n=292,285) | 6.5717 (1.54708) | 6.6246 (1.46356)
  Sleep quantity Change D28(n=292,285) | 0.0015 (1.07390) | -0.0105 (1.10691)
  Sleep quantity Baseline D84(n=285,274) | 6.5456 (1.42402) | 6.6496 (1.34500)
  Sleep quantity Post D84(n=285,274) | 6.5561 (1.43780) | 6.6569 (1.37648)
  Sleep quantity Change D84(n=285,274) | 0.0105 (1.12270) | 0.0073 (1.18906)

16. Secondary Outcome: Summary Statistics of COPD Exacerbations over12 Weeks as Defined by Chronic Pulmonary Disease Tool (EXACT)
Description: The EXACT is a 14-item electronic questionnaire designed to detect the frequency, severity, and duration of exacerbations in patients with COPD.
Time Frame: 12 weeks
Population: Full analysis set consisting of all randomized patients
Measure: Mean (Standard Deviation); unit: COPD exacerbation per participant
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 316 | 313
COPD exacerbation per participant | 0.2 (0.49) | 0.3 (0.56)

17. Secondary Outcome: Time to First COPD Exacerbation
Description: Time-to-event variables will be analyzed by the Kaplan-Meier estimates and the stratified Cox proportional hazard model by smoking status and COPD severity. The model will include treatment and country as factors, and FEV1 prior to inhalation and FEV1 15 min post inhalation of salbutamol/albuterol as covariates. The reported measure will detail the percentage of participants that were event free of a specified event.
Time Frame: 12 weeks
Population: Full analysis set consisting of all randomized patients
Measure: Number (95% Confidence Interval); unit: Percentage of participants event free
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 316 | 313
Percentage of participants event free
  Mild COPD exacerbation | 99.3 [98.4 to 100.0] | 98.7 [97.4 to 100.0]
  Moderate COPD exacerbation | 94.5 [92.0 to 97.1] | 88.5 [84.9 to 92.1]
  Severe COPD exacerbation | 98.0 [96.5 to 99.6] | 98.3 [96.9 to 99.8]
  Moderate or Severe COPD exacerbation | 92.9 [89.9 to 95.7] | 86.8 [82.9 to 90.6]
  Any( mild, moderate,severe) | 92.2 [89.2 to 95.2] | 85.8 [81.9 to 89.8]

18. Secondary Outcome: Annual Rate of COPD Exacerbations
Description: Time-to-event variables will be analyzed by the Kaplan-Meier estimates and the stratified Cox proportional hazard model by smoking status and COPD severity. The model will include treatment and country as factors, and FEV1 prior to inhalation and FEV1 15 min post inhalation of salbutamol/albuterol as covariates.
Time Frame: 12 weeks
Population: Full analysis set consisting of all randomized patients
Measure: Number (95% Confidence Interval); unit: COPD Exacerbations per year
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 316 | 313
COPD Exacerbations per year
  Model based estimates | 0.354 [0.2210 to 0.5663] | 0.659 [0.4523 to 0.9592]
  Actual rate exacerbations per year | 0.39 [NA to NA] — not calculated | 0.73 [NA to NA] — not calculated

19. Secondary Outcome: Duration (in Days) of COPD Exacerbations
Description: Duration and number of the COPD exacerbation will be analyzed by the negative binomial regression model including treatment, country, smoking status, and COPD severity as factors and FEV1 prior to inhalation and FEV1 15 min post inhalation of salbutamol/albuterol as covariates.
Time Frame: 12 weeks
Population: Full analysis set consisting of all randomized patients
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 316 | 313
Days | 1.4 (6.59) | 2.0 (6.28)

20. Secondary Outcome: Percentage of Patients With at Least One Exacerbation up to Week 12
Description: Time-to-event variables will be analyzed by the Kaplan-Meier estimates and the stratified Cox proportional hazard model by smoking status and COPD severity. The model will include treatment and country as factors, and FEV1 prior to inhalation and FEV1 15 min post inhalation of salbutamol/albuterol as covariates. The reported measure will detail the percentage of participants that had an exacerbation up to week 12. Less exacerbations reflect a better outcome.
Time Frame: 12 weeks
Population: Full analysis set consisting of all randomized patients
Measure: Number; unit: Percentage of participants
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 316 | 313
Percentage of participants | 7.6 | 14.1

21. Secondary Outcome: Time (in Days) to Permanent Study Discontinuation Due to COPD Exacerbation
Description: as for outcome 18
Time Frame: 12 weeks
Population: Full analysis set consisting of all randomized patients
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 316 | 313
Days | NA [NA to NA] — number of observations is too small to project time to event | NA [NA to NA] — number of observations is too small to project time to event

22. Secondary Outcome: The Percentage of Patients Who Permanently Discontinued Due to COPD Exacerbation
Description: as for outcome 18
Time Frame: 12 weeks
Population: Full analysis set consisting of all randomized patients
Measure: Number; unit: Percentage participants
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 316 | 313
Percentage participants | 0.6 | 1.6

23. Secondary Outcome: Total Amount (in Doses) of Systemic Corticosteroid Used to Treat COPD Exacerbation During the 12 Week Treatment Period
Description: Total amount (in doses) of systemic corticosteroid used to treat COPD exacerbation will be summarized descriptively by treatment group per each systemic corticosteroid.
Time Frame: 12 weeks
Population: Full analysis set consisting of all randomized patients
Measure: Mean (Standard Deviation); unit: (Prednisolone dose equivalents) mg
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 316 | 313
(Prednisolone dose equivalents) mg
  IM Hydrocortisone (mg) (n=1,0) | 100 (0) | NA (NA) — no participants in this group
  IV dexamethasone (mg) (n=0,1) | NA (NA) — no participants in this group | 4.00 (0)
  IV Hydrocortisone (mg) (n=0,1) | NA (NA) — no participants in this group | 100 (0)
  IV Hydrocortisone sodium succinate (mg) (n=2,0) | 400.00 (282.843) | NA (NA) — no participants in this group
  IV methylprenisolone sodium succinate(mg)(n=1,0) | 250 (0) | NA (NA) — no participants in this group
  IV methylprenisolone sodium succinate(ug)(n=0,1) | NA (NA) — no participants in this group | 80 (0)
  IV prednisolone (mg) (n=0,1) | NA (NA) — no participants in this group | 250 (0)
  Oral Budesonide (mg) (n=0,1) | NA (NA) — no participants in this group | 20 (0)
  Oral methylprenisolone (mg) (n=7,13) | 16.57 (11.414) | 20.31 (9.586)
  Oral prednisolone (mg) (n=8,28) | 24.38 (9.520) | 23.93 (13.060)
  Oral prednisone (mg) (n=8,16) | 31.25 (11.260) | 25.31 (11.176)
  Oral prednisone (ug) (n=0,1) | NA (NA) — no participants in this group | 10 (0)
  Inhalation budesonide (mL)(n=0,1) | NA (NA) — no participants in this group | 0.50 (0)

24. Secondary Outcome: Plasma Cortisol Concentrations at Each Timepoint
Description: Plasma cortisol to be measured in a subset of approximately 60 patients via central laboratory. Blood sample for Plasma cortisol is collected at pre-dose and post dose up to 4 hour on Day 1, up to 12 hours post-dose on Day 28 and Day 84, and 23 hour 35 minute on Day 2, Day 29, and Day 85, and at pre-dose 25 minute on Day 28, and Day 84.
Time Frame: Day 1, Day 28, Day 84
Population: Safety set: A total of 97 (15.4%) patients were included in the 24 h profiling FAS, safety plasma cortisol profiling subgroup, sparse and moderate PK sets.
Measure: Mean (Standard Deviation); unit: nmol/mL
Arm/Group | QMF149 | Salmeterol Xinafoate/Fluticasone Propionate
Number analyzed (Participants) | 50 | 47
nmol/mL
  Baseline (n=45,41) | 328.5 (149.56) | 300.2 (107.36)
  Day 1 / 15 min (n=44,41) | 284.0 (151.96) | 247.1 (91.99)
  Day 1 / 1 hr (n=44,41) | 249.1 (144.90) | 223.0 (85.93)
  Day 1/ 4 hr (n=44,38) | 247.6 (85.90) | 205.7 (68.65)
  Day 1 /23 hr 35 min (n=38,37) | 295.9 (153.80) | 274.2 (115.33)
  Day 28/-25min (n=40,39) | 342.1 (160.16) | 295.6 (98.78)
  Day 28 / 15 min (n=40,39) | 275.0 (140.83) | 239.8 (90.14)
  Day 28 / 1 hr (n=40,39) | 255.9 (134.26) | 211.9 (89.41)
  Day 28 / 4hr (n=40,38) | 241.9 (89.07) | 203.6 (108.62)
  Day 28 / 11hr 35 min (n=40,37) | 124.8 (71.71) | 124.1 (72.39)
  Day 28/ 23 hr 35 min (n=33,32) | 310.6 (99.81) | 306.5 (119.33)
  Day 84 /-25 min (n=41,37) | 337.4 (155.24) | 324.1 (104.01)
  Day 84/ 15 min (n=40,36) | 291.1 (144.26) | 265.5 (103.39)
  Day 84/ 60 min (n=41,38) | 271.3 (158.88) | 236.3 (104.06)
  Day 84/ 4 hr (n=41,38) | 268.4 (136.22) | 224.2 (100.36)
  Day 84/ 11 hr 35 min (n=41,35) | 152.0 (99.66) | 147.5 (108.21)
  Day 84 / 23 hr 35 min (n=37,36) | 339.9 (159.51) | 315.9 (104.67)

25. Secondary Outcome: Plasma Drug Concentrations (Pharmacokinetics) at Each Timepoint
Description: Plasma indacaterol and mometasone furoate is to be measured in a subset of approximately 60 patients via central laboratory. Blood samples are collected at pre-dose on Day 1, 29, and 84; and post dose up to 4 hour on Day 1, up to 12 hours on Day 28 and 84. For sparse pharmacokinetic testing, blood samples will be collected at 23h 35 min post-dose following morning dose administration on Day 28 and 84, in all patients participating in this study.
Time Frame: Day 1, 29, 84
Population: Moderate PK set: A total of 97 (15.4%) patients were included in the 24 h profiling FAS, safety plasma cortisol profiling subgroup, sparse and moderate PK sets.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- QMF149 (Analyte Mometasone Furoate): Assay Analyte: MOMETASONE FUROATE, component of QMF 149 mixture
- QMF149 (Analyte Indacaterol Acetate): Assay Analyte: QAB149 (Indacaterol acetate), component of QMF 149 mixture
Arm/Group | QMF149 (Analyte Mometasone Furoate) | QMF149 (Analyte Indacaterol Acetate)
Number analyzed (Participants) | 50 | 50
pg/mL
  Day 1 time 0 (n=34,44) | 4.17 (13.8) | 4.32 (12.3)
  Day 1 / 15 min (n=44,45) | 31.4 (17.9) | 111 (52.1)
  Day 1 / 1 hr (n=43,45) | 44.6 (19.3) | 89.7 (41.2)
  Day 1/ 4 hr (n=43,45) | 26.8 (15.6) | 51.4 (33.5)
  Day 1 /23 hr 35 min (n=37, 38) | 13.1 (16.7) | 44.8 (69.9)
  Day 28 0 time (n=41,42) | 14.5 (18.0) | 82.0 (47.4)
  Day 28 / 15 min (n= 42,43) | 57.5 (31.6) | 213 (98.0)
  Day 28 / 1 hr (n=41,42) | 68.4 (35.0) | 194 (99.0)
  Day 28 / 4hr (n=42,42) | 43.7 (25.7) | 132 (67.9)
  Day 28 / 11hr 35 min (n=41,42) | 19.2 (12.6) | 86.6 (40.4)
  Day 28/ 23 hr 35 min (n=45,46) | 10.8 (7.32) | 76.5 (38.1)
  Day 84 0 time (n=39,40) | 23.1 (30.5) | 101 (50.8)
  Day 84/ 15 min (n=38,40) | 68.1 (41.4) | 255 (129)
  Day 84/ 60 min (n=38,40) | 84.2 (40.6) | 241 (119)
  Day 84/ 4 hr (n=40,40) | 49.9 (26.4) | 161 (84.6)
  Day 84/ 11 hr 35 min (n=39,41) | 25.9 (21.2) | 115 (67.5)
  Day 84 / 23 hr 35 min (n=44,45) | 14.6 (17.8) | 98.7 (67.8)

26. Secondary Outcome: Pharmacokinetic Parameter: Cmax
Description: Maximum observed plasma concentration after drug administration is to be measured in a subset of approximately 60 patients via central laboratory, and will be determined for indacaterol and MF following morning dosing on Days 28 and 84.
Time Frame: Day 28, 84
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- QMF149 Analyte: Mometasone Furoate: Mometasone furoate as part of QMF149F
- QMF149 Analyte: Indacaterol Acetate: QAB149: indacaterol acetate as a component of QMF149F
Arm/Group | QMF149 Analyte: Mometasone Furoate | QMF149 Analyte: Indacaterol Acetate
Number analyzed (Participants) | 50 | 50
pg/mL
  Day 28 (n=36,35) | 73.3 (24.9) | 215 (71.5)
  Day 84 (n=32,35) | 80.2 (23.0) | 263 (101)

27. Secondary Outcome: Pharmacokinetic Parameter--Tmax
Description: Time to reach the maximum plasma concentration after drug administration is to be measured in a subset of approximately 60 patients via central laboratory, and will be determined for indacaterol and MF following morning dosing on Days 28 and 84.
Time Frame: Day 28, 84
Population: as for outcome 25
Measure: Median (Full Range); unit: Hr
Groups:
- QMF 149 Anaylyte: Mometasone Furorate: Mometasone furoate as a component of QMF149F
Arm/Group | QMF 149 Anaylyte: Mometasone Furorate | QMF149 Analyte: Indacaterol Acetate
Number analyzed (Participants) | 50 | 50
Hr
  Day 28 (n= 36 ,35) | 0.250 (0.833) [0.080 to 3.98] | 0.970 (0.662) [0.230 to 4.15]
  Day 84 (n= 32 ,35) | 0.250 (1.92) [0.220 to 11.7] | 1.00 (1.92) [0.220 to 11.7]

28. Secondary Outcome: Pharmacokinetic Parameter--AUC0-t
Description: Area under the plasma concentration time curve from time zero to time "t" post-dose is to be measured in a subset of approximately 60 patients via central laboratory, and will be determined for indacaterol and MF following morning dosing on Days 28 and 84.
Time Frame: Day 28, 84
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: hr*pg/mL
Groups:
- QMF149 Analyte Mometasone Furoate: QMF149 Mometasone furoate analyte from mixture
- QMF149 Analyte QAB149: QMF149 analyte QAB149 ( indacaterol acetate)
Arm/Group | QMF149 Analyte Mometasone Furoate | QMF149 Analyte QAB149
Number analyzed (Participants) | 50 | 50
hr*pg/mL
  28 Days (n=35,36) | 653 (296) | 2400 (771)
  84 Days (n=31,33) | 693 (297) | 2760 (802)

ADVERSE EVENTS:
Groups:
- SALM/FLUT: SALM/FLUT
Arm/Group | QMF149 | SALM/FLUT
Serious Adverse Events (participants affected / at risk) | 10/316 | 19/313
Other Adverse Events (participants affected / at risk) | 79/316 | 83/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QMF149 (N=316) | SALM/FLUT (N=313)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 2
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
COLITIS (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
MALAISE (General disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1
INCISION SITE INFECTION (Infections and infestations) | 1 | 0
LOBAR PNEUMONIA (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 2 | 0
SPUTUM PURULENT (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
ELECTROCARDIOGRAM T WAVE INVERSION (Investigations) | 0 | 2
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
PLEURAL MESOTHELIOMA MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
INTRACRANIAL ANEURYSM (Nervous system disorders) | 0 | 1
TEMPORAL LOBE EPILEPSY (Nervous system disorders) | 0 | 1
TENSION HEADACHE (Nervous system disorders) | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 0 | 1
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 6 | 5
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QMF149 (N=316) | SALM/FLUT (N=313)
DRY MOUTH (Gastrointestinal disorders) | 4 | 1
NAUSEA (Gastrointestinal disorders) | 4 | 0
FATIGUE (General disorders) | 3 | 4
PYREXIA (General disorders) | 6 | 3
NASOPHARYNGITIS (Infections and infestations) | 12 | 8
RHINITIS (Infections and infestations) | 8 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 4
C-REACTIVE PROTEIN INCREASED (Investigations) | 6 | 2
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 5 | 2
DIZZINESS (Nervous system disorders) | 4 | 0
HEADACHE (Nervous system disorders) | 10 | 5
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 19 | 43
COUGH (Respiratory, thoracic and mediastinal disorders) | 9 | 5
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 | 10
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 6 | 3
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial